CLINICAL TRIAL: NCT00591227
Title: Management of Hyperglycemia in the Emergency Room: A Randomized Clinical Trial of a Subcutaneous Insulin Aspart Protocol Coupled With Rapid Initiation of Basal Bolus Insulin Prior to Hospital Admission Versus Usual Care
Brief Title: Management of Diabetes in the Emergency Room: a Randomized Trial of an Insulin Protocol.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07070902
Record Dates: First submitted 2007-12-27; First posted 2008-01-11 (Estimated); Results first posted 2011-05-05 (Estimated); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Aspart; Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- aspart detemir (Active Comparator): these subjects will be treated with insulin aspart every 2 hours if blood glucose is more than 200 mg/dl during their ER evaluation. If they are admitted to hospital then they will receive a weight-based dose of insulin detemir immediately prior to admission and then every 24 hours thereafter combined with mealtime doses of insulin aspart if they are eating.
  Interventions: Drug: insulin aspart; Drug: insulin detemir
- usual care (No Intervention): these subjects will receive no insulin per protocol during their ER stay or during a possible inpatient admission. The care for their diabetes will be solely determined by the physician(s) in the ER and by the physician(s) caring for them in the hospital if they are admitted. They may receive no therapy, oral agents or insulin per primary physician preference.

INTERVENTIONS:
Drug: insulin aspart — insulin aspart: insulin aspart will be given every 2 hours dosed from 0.05 to 0.15 units per kg weight to patients with a prior history of diabetes if blood glucose is more than 200 mg/dl in the ER.
  If subjects are admitted to hospital then they will receive insulin detemir 0.3 units/kg daily and insulin aspart 0.1 units/kg per meal if they are eating.
  Arms: aspart detemir
Drug: insulin detemir — insulin detemir: insulin aspart will be given every 2 hours dosed from 0.05 to 0.15 units per kg weight to patients with a prior history of diabetes if blood glucose is more than 200 mg/dl in the ER.
  If subjects are admitted to hospital then they will receive insulin detemir 0.3 units/kg daily and insulin aspart 0.1 units/kg per meal if they are eating.If subjects are admitted to hospital then they will receive insulin detemir 0.3 units/kg daily and insulin aspart 0.1 units/kg per meal if they are eating.
  Arms: aspart detemir

SUMMARY:
This study will examine two questions: 1. Whether insulin treatment of high blood sugar in patients with diabetes while they are in the emergency room will improve how quickly they recover from illness if they need to be hospitalized. 2. Whether immediately beginning long lasting insulin detemir in patients with diabetes when they are admitted to hospital from the emergency room will improve how quickly they recover from the illness which necessitated hospitalization.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years
2. History of type 2 diabetes mellitus for at least 3 months
3. Prior therapy with dietary management, oral agents, or insulin
4. Non child-bearing potential or a negative urine pregnancy test
5. Initial blood glucose in ER > 200 mg/dl

Exclusion Criteria:

1. Subsequent finding of diabetic ketoacidosis or hyperosmolar non-ketotic syndrome after initial evaluation.
2. Patients with critical illness suspected to require intensive care unit admission or direct surgical intervention.
3. History of current drug or alcohol abuse.
4. History of current mental illness
5. Inability to give informed consent
6. Female patients who are pregnant or are breast feeding
7. Patients who have clinically significant liver disease with AST/ALT (aspartate transaminase/alanine transaminase) > 3 times the upper range of normal
8. Patients currently treated with dialysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2008-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Baldwin, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Bernard JB, Munoz C, Harper J, Muriello M, Rico E, Baldwin D. Treatment of inpatient hyperglycemia beginning in the emergency department: a randomized trial using insulins aspart and detemir compared with usual care. J Hosp Med. 2011 May;6(5):279-84. doi: 10.1002/jhm.866. PMID 21661100

RESULTS

PARTICIPANT FLOW:
Groups:
- Aspart Detemir: these subjects will be treated with insulin aspart every 2 hours if blood glucose is more than 200 mg/dl during their ER (emergency room) evaluation. If they are admitted to hospital then they will receive a weight-based dose of insulin detemir immediately prior to admission and then every 24 hours thereafter combined with mealtime doses of insulin aspart if they are eating.
Period: Overall Study
Arm/Group | Aspart Detemir | Usual Care
Started | 89 | 87
Completed | 89 | 87
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aspart Detemir | Usual Care | Total
Number analyzed (Participants) | 89 | 87 | 176
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 68 | 68 | 136
  >=65 years | 21 | 19 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (15) | 55 (15) | 55 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 53 | 99
  Male | 43 | 34 | 77
Region of Enrollment [Number; unit: participants]
  United States | 89 | 87 | 176

OUTCOME MEASURES:

1. Primary Outcome: Hospital Length of Stay
Description: hospital length of stay in days
Time Frame: from hospital admission to hospital discharge
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Aspart Detemir | Usual Care
Number analyzed (Participants) | 89 | 87
days | 2.7 [0.7 to 4.7] | 3.1 [1.2 to 5.0]
Statistical Analysis 1: Comparison: Aspart Detemir vs Usual Care; Test type: Superiority or Other; p = 0.58, t-test, 1 sided

2. Secondary Outcome: Average Blood Glucose During the Hospital Admission
Time Frame: from admission to discharge
Population: PI no longer at institution, study is over 10 years old, data unavailable.
Groups:
- Aspart Detemir: these subjects will be treated with insulin aspart every 2 hours if blood glucose is more than 200 mg/dl during their ER evaluation. If they are admitted to hospital then they will receive a weight-based dose of insulin detemir immediately prior to admission and then every 24 hours thereafter combined with mealtime doses of insulin aspart if they are eating.
  insulin aspart: insulin aspart: insulin aspart will be given every 2 hours dosed from 0.05 to 0.15 units per kg weight to patients with a prior history of diabetes if blood glucose is more than 200 mg/dl in the ER.
  If subjects are admitted to hospital then they will receive insulin detemir 0.3 units/kg daily and insulin aspart 0.1 units/kg per meal if they are eating.
  insulin detemir: insulin detemir: insulin aspart will be given every 2 hours dosed from 0.05 to 0.15 units per kg weight to patients with a prior history of diabetes if blood glucose is more than 200 mg/dl in the ER.
  If subjects are admitted to hospital then they will receive insulin detemir 0.3 units/kg daily and insulin aspart 0.1 units/kg per meal if they are eating.If subjects are admitted to hospital then they will receive insulin detemir 0.3 units/kg daily and insulin aspart 0.1 units/kg per meal if they are eating.
Arm/Group | Aspart Detemir | Usual Care
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Frequency of Hypoglycemia
Time Frame: from hospital admission to discharge
Population: PI no longer at institution, study is over 10 years old, data unavailable.
Arm/Group | Aspart Detemir | Usual Care
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Efficacy of Blood Glucose Lowering During the Emergency Room Stay
Time Frame: from emergency room admission to discharge
Population: PI no longer at institution, study is over 10 years old, data unavailable.
Arm/Group | Aspart Detemir | Usual Care
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Frequency of Hypoglycemia During Emergency Room Therapy With Insulin
Time Frame: from emergency room admission to discharge
Population: PI no longer at institution, study is over 10 years old, data unavailable.
Arm/Group | Aspart Detemir | Usual Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Aspart Detemir | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/87
Other Adverse Events (participants affected / at risk) | 0/89 | 0/87

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No